CLINICAL TRIAL: NCT06608875
Title: Precision Sensorimotor Neurorehabilitation Through Personalized Stimulation Loops in a Proof-of-principle Study
Brief Title: Precision Sensorimotor Neurorehabilitation Through Personalized Stimulation Loops
Acronym: StimuLOOP-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Switzerland) (Other); Cereneo AG (Industry); University Children's Hospital, Zurich (Other); Lake Lucerne Institute AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-01400
Record Dates: First submitted 2024-08-09; First posted 2024-09-23 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Consolidation Arm: hyper-personalized feedback based-motor rehabilitation with targeted auditory stimulation during sleep (HPF intervention, TASS intervention)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (participant, care provider, investigator, outcomes assessor).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptation Arm (Sham Comparator): Hyper-personalized feedback-based motor rehabilitation with sham targeted auditory stimulation during sleep (HPF intervention, TASS sham intervention)
  Interventions: Behavioral: Hyper-personalized feedback (HPF intervention); Behavioral: Control targeted auditory stimulation during sleep (TASS sham intervention)
- Consolidation arm (Experimental): Hyper-personalized feedback-based motor rehabilitation with targeted auditory stimulation during sleep (HPF intervention, TASS verum intervention)
  Interventions: Behavioral: Hyper-personalized feedback (HPF intervention); Behavioral: Targeted auditory stimulation during sleep (TASS verum intervention)

INTERVENTIONS:
Behavioral: Hyper-personalized feedback (HPF intervention) — For lower limb motor rehabilitation, the investigator will employ real-time continuous feedback for movement aspects that are specific to each participant's motor deficit. The feedback will be adapted and tailored to each participant.
Behavioral: Targeted auditory stimulation during sleep (TASS verum intervention) — The investigator aim to reactivate rehabilitation- related memories through the presentation of auditory stimuli during sleep with the goal of promoting motor memory consolidation into stable motor commands
  Arms: Consolidation arm
Behavioral: Control targeted auditory stimulation during sleep (TASS sham intervention) — Identical auditory presentation during the motor rehabilitation training, but not during the night (sham promotion memory reactivation)
  Arms: Adaptation Arm

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disease that affects about 1% of the elderly population and accounts for substantial disability and health care costs.

Disability is largely driven by mobility deficits caused by impaired gait. Effective treatments are available to restore lower limb function and improve gait, but response to treatment varies greatly from patient to patient and often shows only small effect sizes. Addressing this heterogeneity requires personalization, a concept referred to precision neurorehabilitation.

StimuLOOP.PD intends to foster structured and reproducible methods for precision neurorehabilitation of gait in PD. The investigator will conduct a proof-of-concept study to investigate a combination of two methods that are each tailored to the individual patient. Two innovative technologies are applied in concert to enhance recovery of lower limb function.

1. Hyper-personalized feedback (HPF): For lower limb motor rehabilitation, the investigator will employ real-time continuous feedback for movement aspects that are specific to each participant's motor deficit. The feedback will be adapted and tailored to each participant. This results in a two-step personalization; in a first step, the investigator will choose what movement aspect is therapeutically targeted, and in a second step, the investigator will define how the feedback is presented to the participant.
2. Targeted auditory stimulation during sleep (TASS):The investigator aim to reactivate rehabilitation- related memories through the presentation of auditory stimuli during sleep with the goal of promoting motor memory consolidation into stable motor commands.

The HPF intervention is expected to induce rapid adaptations, which however do not persist over multiple days. To counter this, the investigator will leverage memory reactivation during sleep to enhance the consolidation of the movement patterns that are learned during HPF.

The investigator expect that these interventions will lead to greater gains in functional walking ability. Beyond demonstrating a proof-of-concept for novel methods of precision neurorehabilitation, positive results of this project may have implications for neurorehabilitation treatment in general by providing first insights into the benefits and interplay of HPF and TASS.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease with gait and postural stability deficits
* ≥18 years of age
* United Parkinson Disease Rating Scale (UPDRS) III gait scores 1-3
* UPDRS III postural instability scores 1-3
* Prescribed rehabilitation therapy at cereneo
* Informed consent as documented by signature
* Adjustments in dopaminergic medication and deep brain stimulation (DBS) to improve motor symptoms implemented to the current best possible extent

Exclusion Criteria:

* Cognitive impairment, Montreal Cognitive Assessment (MoCa) < 20
* Comprehensive aphasia precluding the understanding of study-related information
* Other neurological or medical condition that caused sustained clinically relevant gait and/or postural stability deficits
* Expected acute hospitalization during the training period
* History of a physical or neurological condition that interferes with study procedures
* Social and/or personal circumstances that interfere with the ability to return for therapy sessions and follow-up assessments
* Not capable of voluntary gait adaptation
* Patients taking benzodiazepines or Z-drugs that have a significant effect on sleep EEG
* Recent DBS implant (≤ 6 months)
* Inability to perform outcome assessments without walking aid
* Skin disorders/problems/allergies in face/ear area that could worsen with electrode application (e.g. nickel allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
6 min walking test | Pre, immediately post motor rehabilitation and 1 month post motor rehabilitation
  Change in functional walking ability assessed with the 6 min walking test
MiniBEST test | Pre, immediately post motor rehabilitation and 1 month post motor rehabilitation
  the change in postural stability assessed with the MiniBEST test

SECONDARY OUTCOMES:
Phase Coordination Index | Pre, immediately post motor rehabilitation training and during 15 days of motor rehabilitation training and one-month post-training
  Motor learning assessed via changes in coordination. Coordination assessed using the Phase Coordination Index.
Continuous Relative Phase | Pre, immediately post motor rehabilitation training and during 15 days of motor rehabilitation training and one-month post-training
  Motor learning assessed via changes in coordination. Coordination assessed using Continous Relative Phase.
Variability | Pre, immediately post motor rehabilitation training and during 15 days of motor rehabilitation training and one-month post-training
  Motor learning assessed via changes in variability. Variability assessed using the coefficient of variation (%CV) of common spatio-temporal gait parameters, including stride time, stride length, step length, swing time, stance time, step width, and double limb support time.
Symmetry | Pre, immediately post motor rehabilitation training and during 15 days of motor rehabilitation training and one-month post-training
  Motor learning assessed via changes in symmetry. Symmetry (%) in step length and step time.
Margin of Stability | Pre, immediately post motor rehabilitation training and during 15 days of motor rehabilitation training and one-month post-training
  Motor learning assessed via changes in stability. Stability assessed using Margin of Stability.
Resilience | Pre, immediately post motor rehabilitation training and during 15 days of motor rehabilitation training and one-month post-training
  Motor learning assessed via changes in stability: Stability assessed using resilience metrics.

OTHER OUTCOMES:
Standard sleep architecture measures | During 15 days of motor rehabilitation training
  Single-channel sleep Electroencephalography (EEG): (e.g. % N3, % N2, wake after sleep onset, Sleep efficiency) from scored EEG, electromyography (EMG), and electrooculography (EOG) signal (note: bandpass filtered EMG and EOG signal will only be used for offline sleep scoring according to American Academy of Sleep Medicine standards)
Event related spectral perturbation (ERSP) | During 15 days of motor rehabilitation training
  ERSP: [µV^2/Hz or % or dB of baseline if normalized over time] and event-related potential (ERP) [µV over time] locked to stimuli from frontal, single-channel EEG signal
Frequency spectrum | During 15 days of motor rehabilitation training
  Single-channel sleep EEG: [µV^2/Hz] from frontal, single-channel EEG signal
Slow-wave activity | During 15 days of motor rehabilitation training
  Single-channel sleep EEG: [µV^2/Hz or % or dB of baseline if normalized] in scored non-rapid eye movement (NREM) sleep from frontal, single-channel EEG signal
Sigma power | During 15 days of motor rehabilitation training
  Single-channel sleep EEG: [µV^2/Hz or % or dB of baseline if normalized] in scored NREM sleep from frontal, single-channel EEG signal
Quantity | During 15 days of motor rehabilitation training
  Single-channel sleep EEG: density [number/min], and characteristics (amplitude, peak frequency, bandwidth) of sleep oscillations (spindles, K-complexes, slow-wave-spindle-coupling) in scored NREM sleep from frontal, single-channel EEG signal.
Quality of Life (EQ-5D-5L) | Pre motor rehabilitation training and 1 month after training
  Patient-Reported Outcomes (PRO) measurement that can assess patients' quality of life, irrespective of the disease.
  Quality of life scale developed by EuroQol Group called EQ-5D-5L, scoring from level 1 indicating no problem to level 5 indicating extreme problems.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No